CLINICAL TRIAL: NCT06315218
Title: Examining the Health Effects of iTHRIVE 365 Among Black Same Gender Loving Men
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Positive Impact Health Centers (Other); George Washington University (Other); Carnegie Mellon University (Other); Emory University (Other); Columbia University (Other); Arizona State University (Other); Thrive Social Services (Other)
Responsible Party: Principal Investigator, Devin English, PhD, Devin English, PhD; Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro2023000968
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Sexual and Gender Minorities; Social Stigma; Medication Adherence; Depressive Symptoms; Anxiety Symptoms
MeSH Terms: conditions — Coitus; Social Stigma; Medication Adherence; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): iTHRIVE 365 is a multicomponent intervention that combines mHealth features and institutional to support community priorities identified in formative CBPR. In line with best-practices for trials of intervention principles (TIPs) with mHealth interventions, iTHRIVE 365 deploys intervention elements that serve to accomplish intervention strategies. iTHRIVE 365 intervention strategies are to promote: 1)Health knowledge and motivation; 2)Social support coping; 3)Access to culturally-affirming healthcare; and 4)Housing and other economic resources. iTHRIVE 365 pursues these strategies via these intervention elements: 1)Weekly HIV and psychological health information and motivation content and daily health notifications; 2)Online moderated forums, interpersonal chats, and community calendars; 3)Linkage to biopsychosocial healthcare via THRIVE SS's network of Black SGLM-affirming providers; and 4)Housing and economic resources through THRIVE SS's direct support and referral network.
  Interventions: Behavioral: iTHRIVE 365 HIV care intervention
- Control Arm (No Intervention): The 6-month waitlist control group will only have access to THRIVE SS services not encompassed by iTHRIVE 365, such as in-person events. The investigators will ensure the control group does not access the iTHRIVE 365 mHealth app portion by screening all new app users, giving the intervention group unique private log-ins, and explaining the importance of securing those log-ins to ensure the accuracy of study results.

INTERVENTIONS:
Behavioral: iTHRIVE 365 HIV care intervention — iTHRIVE 365 is a multicomponent intervention that combines mHealth features and institutional to support community priorities identified in formative CBPR. In line with best-practices for trials of intervention principles (TIPs) with mHealth interventions, iTHRIVE 365 deploys intervention elements that serve to accomplish intervention strategies. iTHRIVE 365 intervention strategies are to promote: 1)Health knowledge and motivation; 2)Social support coping; 3)Access to culturally-affirming healthcare; and 4)Housing and other economic resources. iTHRIVE 365 pursues these strategies via these intervention elements: 1)Weekly HIV and psychological health information and motivation content and daily health notifications; 2)Online moderated forums, interpersonal chats, and community calendars; 3)Linkage to biopsychosocial healthcare via THRIVE SS's network of Black SGLM-affirming providers; and 4)Housing and economic resources through THRIVE SS's direct support and referral network.
  Arms: Intervention Arm

SUMMARY:
This research study aims to test the effectiveness, reach, and maintenance over time of the iTHRIVE 365 intervention for Black same gender loving men (SGLM) living with HIV. iTHRIVE 365 is a SGLM community-developed multicomponent mHealth intervention that aims to: 1) Support daily health promotion via HIV and psychological health education and health maintenance reminders; 2) Foster positive social connections among SGLM via online moderated forums, interpersonal chats, and community calendars; 3) Connect clients to SGLM-affirming healthcare, including HIV treatment and mental healthcare; 4) Provide resources for housing, transportation, and other economic empowerment.

DETAILED DESCRIPTION:
This research study aims to test the effectiveness, reach, and maintenance over time of the iTHRIVE 365 intervention for Black same-gender loving men (SGLM) living with HIV. I thrive 365 is an SGLM community-developed multicomponent intervention that aims to: 1) Support daily health promotion via HIV and psychological health education and health maintenance reminders; 2) Foster positive social connections among SGLM via online moderated forums, interpersonal chats, and community calendars; 3) Connect clients to SGLM-affirming healthcare, including HIV treatment and mental healthcare; 4) Provide resources for housing, transportation, and other economic empowerment.

The investigators will pursue the following aims:

1. Test the effectiveness of THRIVE365 in improving daily and longer-term (1-6 months) HIV-related behavioral health (primary outcome: ART adherence) and psychological health (e.g., secondary outcomes: lower depressive and anxiety symptoms) in a 6-month waitlist randomized controlled trial with 350 Black SGLM living with HIV in the four Atlanta-area Ending the HIV Epidemic (EHE) jurisdictions.
2. Examine the moderating effect of THRIVE365 on associations between intersectional stigma (e.g., intersectional racist, heterosexist, and HIV stigma) and our primary and secondary HIV outcomes.
3. Evaluate THRIVE365 maintenance and reach the user level (e.g., within-user changes in engagement and daily effects) and setting level (e.g., intervention adaptations, Black SGLM community uptake).

Participants will be recruited in collaboration with THRIVE SS, the most prominent Black SGLM-led social service organization for Black SGLM in the Atlanta, GA metro area. After completing an online screener to assess basic eligibility requirements, participants will be scheduled for an online Health Insurance Portability and Accountability Act (HIPPA)---compliant Zoom consent and baseline survey process. All online assessments will be completed using HIPAA-compliant Qualtrics surveys. Participants will review study information and complete informed consent procedures with study staff, including agreeing to provide access to their iTHRIVE 365 paradata and HIV viral suppression results. Once consented, participants will complete a computerized retrospective interview to assess HIV anti-retroviral treatment (ART) adherence and substance use, as well as measures of intersectional stigma, depressive symptoms, anxiety symptoms, emotion regulation, social support coping, ART information and motivation, and multilevel barriers to ART adherence. Participants will also be guided through a practice daily diary. Finally, intervention group participants will be registered for the mHealth (e.g., online forums) and institutional (e.g., linkage to care) aspects of iTHRIVE 365. Control group participants will remain on the registration waitlist until after the 6-month study is over. All participants will receive virtual gift card compensation directly following the baseline.

All participants will complete brief daily measures of intersectional stigma, ART adherence, substance use, depressive and anxiety symptoms, emotion regulation, and social support coping for 14 days after baseline to assess daily iTHRIVE 365 effectiveness. Upon completing the 2-week cycle, participants will complete a 2-week follow-up online survey, including identical measures to those received at baseline. All participants will receive compensation for their participation in the 2-week assessment and compensation based on the number of daily surveys the participants completed.

There will be online follow-up surveys at 1-, 2-, 4-, and 6-months post baseline. These assessments will include measures identical to the baseline and 2-week assessments. As with the baseline, participants will receive virtual gift card compensation directly after participants complete their surveys. Following the 6-month assessment, all participants will participate in a second 2-week daily diary study. At the end of the 2-week process, participants will engage in a debriefing session and be able to provide feedback on the iTHRIVE 365 intervention and the research process. As with the initial daily diary period, participants will receive virtual gift card compensation based on the number of surveys completed.

To accomplish study aims, the investigators will estimate all analytic models in Mplus and SPSS. The investigators will test the effectiveness of iTHRIVE 365 on daily primary and secondary HIV and psychological outcomes by examining a series of two-level dynamic structural equation models (DSEMs) that test differences in within-participant changes in our outcomes across intervention groups. The investigators will test the effectiveness of iTHRIVE 365 on longer-term primary and secondary outcomes through between- and within-group analyses estimated as latent growth curve models that test changes in the outcomes across intervention groups during the 6-month study period. The investigators will examine the main effects of intersectional stigma on primary and secondary outcomes using DSEM in autoregressive models (VAR (1)). The investigators will build off these VAR (1) models to examine the moderating effects of iTHRIVE 365 on the intersectional stigma HIV outcomes associations using multiple group moderation analyses. The investigators will run all descriptive analyses in SPSS for reach and maintenance. Effects maintenance analyses will build off the DSEM and VAR (1) models to observe time as a predictor of changes within and across participants in the iTHRIVE 365 effects.

ELIGIBILITY:
Inclusion Criteria:

1. Identify as Black or African American, regardless of ethnicity
2. Identify as male, regardless of sex assigned at birth
3. Are living with HIV and prescribed a daily ART regimen
4. Are age ≥ 18;
5. Have sex with men
6. Own an internet-connected device (e.g., smartphone, tablet)
7. Reside in the Atlanta-area EHE jurisdictions.

Exclusion Criteria:

1. Lack of English fluency
2. Past participation in the pilot.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Anyone that identifies as a man.
Enrollment: 350 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Antiretroviral (ART) Medication Use | 24 hours
  For daily surveys, participants will report ART adherence on a single binary item ("In the past 24 hours did the participant take ART medication?")
ART adherence-Long Lag Assessments | 2 weeks
  The investigators will use the NAME scale that assesses barriers to ART adherence.

SECONDARY OUTCOMES:
Daily Diary Substance Use | 24 hours
  The investigators will measure daily substance use with single-item binary measures of various substances (e.g.,alcohol, marijuana).
Substance Use-Long Lag Assessments | 2 weeks
  For long lags (i.e., 2 week assessment to 6 month assessment), participants will complete an online, automated retrospective assessment of substance use in the past 2 weeks.
Depressive Symptoms | 24 hours
  The Patient Health Questionnaire-4 assesses anxiety and depressive symptoms. Participants rate the extent to which the participants had been experiencing each item the past day (e.g., "In the past 24 hours, I've been feeling nervous, anxious, or on edge") on a scale from 0 (not at all) to 3 (entirely). The investigators used an average across all items for each time point.
Depressive Symptoms-Long Lag | 2 weeks
  The Brief Symptom Inventory assesses anxiety and depressive symptoms. Participants rate the extent to which the participants had been experiencing each item the past two weeks (e.g., "Feeling hopeless about the future") on a scale from 0 (not at all) to 4 (Extremely). The investigators will use an average across all items for each time point.
Anxiety Symptoms | 24 hours
  The Patient Health Questionnaire-4 assesses anxiety and depressive symptoms. Participants rate the extent to which the participants had been experiencing each item the past day (e.g., "In the past 24 hours, I've been feeling nervous, anxious, or on edge") on a scale from 0 (not at all) to 3 (completely). We used an average across all items for each time point.
Anxiety Symptoms-Long Lag | 2 weeks
  The Brief Symptom Inventory assesses anxiety and depressive symptoms. Participants rate the extent to which the participants had been experiencing each item the past 2 weeks (e.g., "Feeling tense or keyed up") on a scale from 0 (not at all) to 4 (Extremely). The investigators will use an average across all items for each time point.
Emotion Regulation Emotion Regulation | 24 hours
  A validated four-item version of the Difficulties with Emotion Regulation Scale assesses emotion regulation. Participants rated the extent to which the participants had been experiencing each item (e.g., "In the past 24 hours, I've been experiencing my emotions as overwhelming") in the past day on a scale from 0 (not at all) to 3 (entirely). The investigators used an average across all items for each time point.
Emotion Regulation-Long Lag Assessments | 2 weeks
  The investigators will use the Difficulties with Emotion Regulation Scale- Short Form (DERS-SF) for long lags
COPE | 24 hours
  A modified version of the Brief-COPE assesses coping approaches to stress over the last 24 hour. It includes the 6 items from the interconnectedness and problem-oriented subscales, and 3 original items assessing specific interconnectedness with Black LGBTQ people and problem-oriented action against injustice.
COPE-Long Lag Assessments | 2 weeks
  The investigators will use the Brief-COPE measure to assess past 2-week coping, which assesses the following coping approaches in 28 items: Self-distraction, active coping, denial, substance use, use of emotional social support, use of instrumental social support, Behavioral disengagement, venting, positive reframing, planning, humor, acceptance, religion, and self-blame.

CONTACTS AND LOCATIONS:
Overall Officials: Devin English, Ph.D., Principal Investigator — Rutgers University; Justin Smith, MS, MPH, Principal Investigator — Positive Impact Health Centers

IPD SHARING:
Plan to Share IPD: Yes
Outside researchers will be able to request access to these de-identified data through email to the PI in order to conduct analyses for which the PI and study team do not have expertise. This request will be considered by the PI, the appropriate officers at Rutgers University for processing. As such, the PI will initiate a DTA, and seek the legal advice of Rutgers University regarding the adequacy of compliance with any relevant laws, policies, or regulations. If approved, data will be completely de-identified and shared through a secure sharing mechanism (e.g., password protected and encrypted online database for electronic data). No participant codes will be shared with external researchers.
Supporting Information: Study Protocol, SAP
Time Frame: Data will only be shared with other researchers who have received IRB approval and who will destroy or return dataset information after completing their analyses.
Access Criteria: Data will only be shared with other researchers who have received IRB approval and who will destroy or return dataset information after completing their analyses.

REFERENCES:
- [Background] English D, Smith JC, Scott-Walker L, Lopez FG, Morris M, Reid M, Lashay C, Bridges D, McNeish D. Feasibility, Acceptability, and Preliminary HIV Care and Psychological Health Effects of iTHRIVE 365 for Black Same Gender Loving Men. J Acquir Immune Defic Syndr. 2023 May 1;93(1):55-63. doi: 10.1097/QAI.0000000000003167. PMID 36706362
- [Background] English D, Smith JC, Scott-Walker L, Lopez FG, Morris M, Reid M, Lashay C, Bridges D, Rosales A, Cunningham DJ. iTHRIVE 365: A Community-Led, Multicomponent Health Promotion Intervention for Black Same Gender Loving Men. Ann LGBTQ Public Popul Health. 2023 Dec;4(4):363-383. doi: 10.1891/lgbtq-2022-0009. PMID 39055282
- See also: iTHRIVE 365: A Community-Led, Multicomponent Health Promotion Intervention for Black Same Gender Loving Men — https://connect.springerpub.com/content/sgrlgbtq/early/2023/05/09/lgbtq-2022-0009